CLINICAL TRIAL: NCT05349032
Title: Assessing the Bioavailability of Leading Phytonutrient Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epiceutical Labs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 101
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Inflammation
Keywords: infalmmation; bioavailability
MeSH Terms: conditions — Inflammation | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Meriva (Other): 120 mg of curcumin in Meriva.
  Interventions: Dietary Supplement: Curcumin
- Longvida (Other): 120 mg of curcumin Longvida.
  Interventions: Dietary Supplement: Curcumin
- NovaSol (Other): 120 mg of curcumin NovaSol
  Interventions: Dietary Supplement: Curcumin
- CurcElite (Other): 120 mg of curcumin CurcElite
  Interventions: Dietary Supplement: Curcumin
- UltaCur (Other): 120 mg of curcumin Ultracur
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — Oral supplement

SUMMARY:
This study will primarily test various phytonutrient-based supplements to see which gets absorbed into the body the best. The study will secondarily look at inflammatory markers in the urine to determine any change.

DETAILED DESCRIPTION:
This study will primarily test various phytonutrient-based supplements to see which gets absorbed into the body the best. 120 mg of curcumin from brands Meriva, CurcElite, Lonvida, UltraCur, NovaSol. The study will secondarily look at inflammatory markers in the urine to determine any change.

ELIGIBILITY:
Inclusion Criteria:

* Age and gender

Exclusion Criteria:

* Cannot take any phytonutrient or curcumin supplement five days prior to commencement.

Ages: 21 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Bioavailability | 0, 1, 2, 4, and 12 hours
  Blood Plasma

CONTACTS AND LOCATIONS:
Locations (1):
- David Roberts, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Blood plasma and urine samples will be collected for five different times over five different supplements.

REFERENCES:
- [Result] Jamwal R. Bioavailable curcumin formulations: A review of pharmacokinetic studies in healthy volunteers. J Integr Med. 2018 Nov;16(6):367-374. doi: 10.1016/j.joim.2018.07.001. Epub 2018 Jul 4. PMID 30006023